CLINICAL TRIAL: NCT00665613
Title: The Relationship Between Osteoporosis and Chronic Oral Anticoagulation Therapy With Warfarin
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Mario Castellanos, Clinical Director of Research for Dept. of Medicine, Northwell Health
Other Study IDs: 04-054
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Osteoporosis
Keywords: warfarin use
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine if osteoporosis is an unrecognized complication of chronic anticoagulation with warfarin.

ELIGIBILITY:
Inclusion Criteria:

* Patients on warfarin that have had BMD within a year

Exclusion Criteria:

* Patients on bisphosphates, SERMS, anticonvulsants, estrogens, androgens, calcitonin, hctz and thyroid hormone replacement

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients on warfarintherapy in the SIUH coumadin center
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2004-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Bone Density | 5 to 10 years
  bone density as measured by xray to assess bone strength nd risk of fracture

CONTACTS AND LOCATIONS:
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States